CLINICAL TRIAL: NCT06697808
Title: Cranial Ultrasound for Point of Care Intracranial Pathology Detection in Pediatrics (CUPID-Peds)
Brief Title: Cranial Ultrasound for Point of Care Intracranial Pathology Detection in Pediatrics
Acronym: CUPID-Peds
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00111568
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury
Keywords: head injury; imaging; pediatrics
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To improve patient selection for head CT, a safe and high sensitivity screening neuroimaging modality is needed. Currently many clinicians must make treatment decisions based solely on the patients clinical exam, which has low sensitivity and specificity and low inter-rater reliability. This study is being done to learn more about B-mode cranial point-of-care ultrasound (cPOCUS). Ultrasound has several advantages. It is a safe, non- invasive, low-cost, fast and portable bedside tool without ionizing radiation exposure.

DETAILED DESCRIPTION:
B-mode cranial point-of-care ultrasound (cPOCUS) being used in this study is an innovative, low-risk, inexpensive solution for diagnosing clinically significant intracranial pathology in children presenting with blunt head trauma which could be valuable for resource- austere environments. Traumatic brain injury remains a leading cause of death and disability in children. In addition, those who present with suspected acute brain injury in resource-austere environments may be at high risk of long-term neurologic sequelae or death. Early neuroimaging to identify traumatic brain injury and guide interventions is key to preventing their neurologic morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a head computed tomography (CT) as the standard of care
* Seen in the pediatric Emergency Department or Pediatric Intensive Care Unit at Atrium Health Wake Forest Brenner Children's Hospital or Levine Children's Hospital

Exclusion Criteria:

* Patients with open skull fractures
* Previous hemicraniectomy
* Existing surgical defect in the skull
* Patients being transitioned to comfort care

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients in the Emergency Department or Pediatric Intensive Care Unit due blunt head trauma.
Sampling Method: Probability Sample
Enrollment: 169 (Estimated)
Dates: Start 2024-11-24 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Cranial Point-of-Care Ultrasound | Day 1
  The diagnostic accuracy of cranial point-of-care ultrasound (cPOCUS) is reported reported by comparing the counts of positive and negative findings for the two imaging modalities with sensitivity, specificity, positive predictive value and negative predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Fraga, MD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No